CLINICAL TRIAL: NCT01564017
Title: Phase II, Multicenter, Randomized, Double-blind Study, With Subcutaneous Immunotherapy, in Parallel Groups and Placebo-controlled, in Patients With Rhinoconjunctivitis ± Asthma Sensitized to Dermatophagoides Pteronyssinus.
Brief Title: Dose-response Study With Subcutaneous Immunotherapy of an Standardized Dermatophagoides Pteronyssinus (DPT) Extract
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Roxall Medicina España S.A (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BIA--DPT-P2-001; 2011-004583-30 (EudraCT Number)
Record Dates: First submitted 2012-03-23; First posted 2012-03-27 (Estimated); Last update posted 2017-05-01 (Actual); Status verified 2017-04

CONDITIONS: Allergic Rhinoconjunctivitis
Keywords: Allergy; Allergic rhinoconjunctivitis; Immunotherapy; D. pteronyssinus; house dust allergy
MeSH Terms: conditions — Hypersensitivity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- Allergovac depot. Group 1 (Experimental): Increasing dosages till the maintenance dose of 0.0625 SPT is reached. Afterwards, 3 maintenance doses are given at 4-weekly intervals.
  Interventions: Biological: Allergovac depot
- Allergovac depot. Group 2 (Experimental): Increasing dosages till the maintenance dose of 0.125 SPT is reached. Afterwards, 3 maintenance doses are given at 4-weekly intervals.
  Interventions: Biological: Allergovac depot
- Allergovac depot. Group 3 (Experimental): Increasing dosages till the maintenance dose of 0.25 SPT is reached. Afterwards, 3 maintenance doses are given at 4-weekly intervals.
  Interventions: Biological: Allergovac depot
- Allergovac depot. Group 4 (Experimental): Increasing dosages till the maintenance dose of 0.5 SPT is reached. Afterwards, 3 maintenance doses are given at 4-weekly intervals.
  Interventions: Biological: Allergovac depot
- Allergovac depot. Group 5 (Experimental): Increasing dosages till the maintenance dose of 0.75 SPT is reached. Afterwards, 3 maintenance doses are given at 4-weekly intervals.
  Interventions: Biological: Allergovac depot
- Allergovac depot placebo. Group 6 (Placebo Comparator): The same scheme of treatment as the active groups
  Interventions: Biological: Allergovac depot

INTERVENTIONS:
Biological: Allergovac depot — Depot sterile suspension fpor subcutaneous injection
  Increasing concentrations to reach the following maintenance doses:
  Group 1: 0.25 SPT
  Arms: Allergovac depot. Group 1
Biological: Allergovac depot — Depot sterile suspension for subcutaneous injection.
  Increasing concentrations to reach the following maintenance doses:
  Group 2: 0.5 SPT
  Arms: Allergovac depot. Group 2
Biological: Allergovac depot — Depot sterile suspension for subcutaneous injection.
  Increasing concentrations to reach the following maintenance doses:
  Group 3: 1 SPT
  Arms: Allergovac depot. Group 3
Biological: Allergovac depot — depot sterile suspension for subcutaneous injection
  Increasing concentrations to reach the following maintenance doses:
  Group 4: 2 SPT
  Arms: Allergovac depot. Group 4
Biological: Allergovac depot — Depot sterile suspension for subcutaneous injection.
  Increasing concentrations to reach the following maintenance doses:
  Group 5: 4 SPT
  Arms: Allergovac depot. Group 5
Biological: Allergovac depot — Sterile suspension for subcutaneous injection.
  Same number of administration as the active groups
  Arms: Allergovac depot placebo. Group 6

SUMMARY:
As part of the registration plan of our products and after performing a Phase I study the present trial has been designed to compare the efficacy of 5 different doses of subcutaneous immunotherapy in depot presentation.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must sign the Informed Consent Form.
2. Patients must be between 18 and 60 years of age.
3. Patients with perennial allergic rhinoconjunctivitis produced by Dermatophagoides pteronyssinus during at least 2 years prior to participating in the study. Although the pathology being studied is allergic rhinoconjunctivitis, patients who have concomitant mild or moderate asthma may be included.
4. Patients who have had a skin prick test result greater or equal to 3 mm in diameter against Dermatophagoides pteronyssinus.
5. Patients who have specific Immunoglobulin E (IgE) greater or equal to class 2 (CAP/PHADIA) to Dermatophagoides pteronyssinus.
6. Patients will preferably be monosensitized to Dermatophagoides pteronyssinus. Polysensitized patients may only be included in the study if their other sensitizations are produced by:

   * Pollens whose season period does not overlap with the study treatment or, if overlap, whose specific IgE levels are less than class 2.
   * Perennial allergens with specific IgE levels less than class 2.
   * Allergens that do not cohabit with the patient or whose environmental levels are not high enough to produce symptoms during the study period.
7. Women of child-bearing potential must have a negative urine pregnancy test at the time they begin the study.
8. Furthermore, women of child-bearing potential must agree to use adequate contraceptive methods during this study if they are sexually active.

Exclusion Criteria:

1. Patients with stable and continued use of medication to treat their allergic condition during the 2 weeks prior to their inclusion in the study.
2. Patients sensitized and with specific IgE levels greater or equal to class 2 to other perennial or seasonal allergens clinically relevant including other mites unless they are cross reactive with Dermatophagoides pteronyssinus.
3. Patients who have received immunotherapy in the 5 years prior to the study against either the allergen being tested or an allergen which is cross-reactive, or who are currently receiving immunotherapy for any other allergen.
4. Patients with severe asthma or FEV1< 70% or with asthma which requires treatment with inhaled or systemic corticoids at the time of the study or in the 8 weeks immediately prior to the onset of treatment.
5. Patients with immunological, cardiac, renal or hepatic diseases or with any other illness which the investigators deem may interfere with the study.
6. Patients with a prior history of anaphylaxis.
7. Patients with chronic urticaria.
8. Patients with moderate-severe atopic dermatitis.
9. Patients with clinically relevant malformations of the upper respiratory tract.
10. Patients who have participated in another clinical trial within 3 months prior to this study.
11. Patients being treated with tricyclic antidepressants, psychotropic drugs, beta-blockers, or angiotensin-converting enzyme inhibitors (ACEIs).
12. Women who are pregnant or breast-feeding or are of child-bearing age and who do not agree to use adequate contraception if they are sexually active and who have not demonstrated that they have been surgically sterilized or have other means of not bearing children.
13. Patients who cannot attend study visits.
14. Patients who are uncooperative or refuse to participate in the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2012-05; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Changes in nasal provocation test | from baseline (V0) to final visit (VF 18 weeks after randmization)
  Variation of the concentration of DPT extract needed to produce a positive nasal provocation test from baseline (V0) to final visit (FV). The changes will be compared among groups (including the placebo group).

CONTACTS AND LOCATIONS:
Overall Officials: Fernando Rodríguez, MD, Principal Investigator — Hospital Universitario Marqués de Valdecilla; Ramón Lleonart, MD, Principal Investigator — Hospital Universitario Marqués de Valdecilla; Albert Roger, MD, Principal Investigator — Germans Trias i Pujol Hospital; Dolores Hernández, MD, Principal Investigator — Hospital Universitario La Fe; Carmen Vidal, MD, Principal Investigator — Complejo Hospitalario Universitario de Santiago; Juan A Pagán, MD, Principal Investigator — Hospital Virgen de la Arrixaca; Carmen Marcos, MD, Principal Investigator — Hospital Xeral de Vigo; Jose A Navarro, MD, Principal Investigator — Hospital Donostia; Victoria Moreno, MD, Principal Investigator — Hospital Blanca Paloma; Luis A Navarro, MD, Principal Investigator — Hospital Luis Alcañiz; María I Peña, MD, Principal Investigator — Hospital Vega Baja; Marta Alvariño, MD, Principal Investigator — Hospital de Manises
Locations (12):
- Spain (12):
  - Hospital Vega Baja, Orihuela, Alicante
  - Hospital Germans Triasl i Pujol, Badalona, Barcelona
  - Hospital Donostia, Donostia / San Sebastian, Guipuzcoa
  - Complejo Hospitalario Universitario de Santiago, Santiago de Compostela, La Coruña
  - Hospital Virgen de la Arrixaca, El Palmar, Murcia
  - Hospital Xeral de Vigo, Vigo, Pontevedra
  - Hospital de Manises, Manises, Valencia
  - Hospital Luis Alcañiz, Xátiva, Valencia
  - Hospital Universitari de Bellvitge, Barcelona
  - Hospital Blanca Paloma, Huelva
  - Hospital Marqués de Valdecilla, Santander
  - Hospital Universitari i Politècnic La Fe, Valencia